CLINICAL TRIAL: NCT00732511
Title: Effect of Coreg CR on BP, Endothelial Function, Exhaled Nitric Oxide, and Nitric Oxide Production and Oxidation
Brief Title: Coreg CR, Blood Vessel Stiffness and Blood Vessel Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Nathaniel Winer, M.D., Principal Investigator, State University of New York Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Glaxo Smith Kline 111105
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Endothelial Function; Diabetes Mellitus; Hypertension
Keywords: Endothelial dysfunction; Blood vessel stiffness; Nitric oxide; Oxidative stress
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Coreg Cr will be up-titrated as needed to achieve blood pressure <130/80
  Interventions: Drug: carvedilol
- 2 (Active Comparator): Toprol XL will be up-titrated at weekly intervals to achieve a blood pressure <130/80 mm Hg
  Interventions: Drug: metoprolol extended release

INTERVENTIONS:
Drug: carvedilol — capsules in doses of 20, 40, and 80 mg; once daily; 12 weeks duration
  Other Names: Coreg CR
  Arms: 1
Drug: metoprolol extended release — tablets in doses 50, 100, and 200 mg; once daily; 12 weeks duration
  Other Names: Toprol XL
  Arms: 2

SUMMARY:
We are comparing the blood pressure-lowering effects of two marketed medications, Coreg CR and Toprol XL. Although both drugs reduce blood pressure by blocking the action of noradrenaline on beta-receptors in the blood vessels, Coreg CR also blocks alpha-receptors, which may provide added blood pressure-lowering. In addition, Coreg CR may have anti-oxidant actions. Cells which line blood vessels (termed "endothelial cells") make nitric oxide (NO), which relaxes the muscle cells encircling the blood vessels, causing a reduction in blood pressure. When body cells use oxygen, they normally produce "free radicals", which can destroy NO,leading to high blood pressure, heart damage and worsenimg of diabetes. Antioxidants remove free radicals and prevent or repair this damage. In this study we will measure endothelial cell function, blood vessel wall stiffness, NO in exhaled breath, and blood levels of substances which reflect NO production and destruction to determine if a pure beta-blocker (Toprol XL) differs from an alpha/beta blocker (Coreg CR) in these effects. We will also examine the mechanism by which such differences might occur.

DETAILED DESCRIPTION:
The following techniques will be used:

Endothelial function will be measured non-invasively by flow-mediated changes in pulsatile blood volume in the finger-tips.

Vascular compliance (stiffness) will be assessed by tonometry of the radial pulse wave ("augmentation index") and diastolic puse wave analysis.

Plasma nitrate/nitrite levels mirror NO production and will be measured spectrophotometrically by the Griess reaction.

Plasma nitrotyrosine, an in vivo marker of NO-dependent damage induced by reactive nitrogen intermediates derived from NO, will be measured by ELISA.

Exhaled NO may provide an real-time measure of endothelial cell NO production and can be measured by a hand-held device which contains an electrochemical detector sensitive to 5 ppb.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus,
2. Stable antidiabetic regimen for 3 months
3. Hemoglobin A1c <8.6%
4. Stable antihypertensive medication regimen for 3 months or more, including either an angiotensin-converting enzyme inhibitor or angiotensin receptor blocker

Exclusion Criteria:

1. Any clinically significant abnormality on history, physical examination, or laboratory testing which could preclude safe completion of the study
2. Significant cardiac conditions
3. Lung disease
4. Cigarette smoking
5. Chronic kidney disease (Stage 3 or greater)
6. Type 1 diabetes
7. Known contraindication to alpha- or beta-blocker therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-12 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Effect of Coreg CR compared to Toprol XL on endothelial function, vascular compliance, and parameters of oxidative stress from time of randomization to study drug termination | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Winer, M.D., Principal Investigator — Stae University of New York Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States